CLINICAL TRIAL: NCT00189618
Title: The Effects of Physical Training, Aspirin, and Clopidogrel on the Walking Capacity of Patients With Stage II Peripheral Arterial Disease
Brief Title: The Effects of Physical Training, ASA (Aspirin), and Clopidogrel on the Walking Capacity of Patients With Stage II Peripheral Arterial Disease (PAD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arteriogenesis Competence Network (Other)
Responsible Party: PD Dr. K.-H. Labs, Arteriogenesis Competence Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AN0104
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral vascular disease; Peripheral arterial disease; Walking Capacity; Aspirin; Clopidogrel
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Aspirin
- 2 (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Aspirin — 100mg p.o. OD
  Arms: 1
Drug: Clopidogrel — 75mg p.o. OD
  Arms: 2

SUMMARY:
To evaluate the change in walking capacity after a well organized and structured intensive physical training program with supportive pharmacotherapy with Clopidogrel or ASA. It is hypothesized that statistically superior results will emerge from a structured training supported by Clopidogrel as compared to a structured training supported by ASA.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) can not be seen in isolation but represents the peripheral manifestation of a generalized atherosclerosis. The co-morbidity with coronary heart disease and/or a cerebral atherosclerosis ranges between 20 % and 90 %, depending on the degree of severity of PAD from 1-5. The relative risk of a (predominantly cardiac) death is increased by a factor of 2 already in asymptomatic PAD patients; the risk will increase furthermore by another factor of 2 to 4 when patients become symptomatic. PAD is not a rare disease but has a prevalence of 15 % to 20 % in an elderly western population (> 50 years of age). While the clinical presentation of PAD is relatively benign in the majority of cases, the disease carries a high risk potential with high directly and indirectly related costs. Thus, from a medical but also from a socio-economic point of view, there is the need to control the PAD complication rate and related treatment costs as effectively as possible.

The most physiological treatment approach, which is internationally accepted, is physical training. There is agreement, that physical training does improve the collateralisation of vascular lesions, does improve the rheologic properties of blood, but does also lead to a shift from glycolytic (type 2) to oxidative (type 1) muscle fibers in the working musculature. This shift is associated with an increase in capillary density, a fact which subsequently favors an optimal oxygen extraction and oxygen utilisation. Another effect of physical training, which may be of utmost importance, relates to its potential to modify the patients risk factor profile. It was shown in epidemiological, clinical, and experimental studies, that even a moderate physical training does increase the insulin receptor sensitivity (and hence positively influences one of the major factors for atherosclerosis), does increase the fibrinolytic activity following prothrombotic stimulation, does decrease the diastolic blood pressure in hypertensive patients, does decrease the LDL/HDL ratio, and does decrease the overall cardiac mortality.

The aim of any treatment of intermittent claudication is a clinically relevant improvement in the patient's mobility and quality-of-life. In a previous study it was shown, that a 3 months structured, supervised PAD rehabilitation program will satisfy this demand and will lead to an improvement of the initial (painfree) claudication distance of approximately 190%. One third of the patients of this study were started on Clopidogrel as a supportive pharmacotherapy at the beginning of the trial. It was interesting to note that optimal training results (defined as an improvement of the ICD by > 200 %) were only seen in patients who were treated with Clopidogrel but were not reported from patients who received ASA (aspirin) on top of training.

Non-published data from the Art.Net. preclinical group (Dr. I. Höfer, Dr. I. Buschmann, Freiburg), which were presented at an Art.Net. meeting on March 24, 2003 showed that using a rabbit hind leg model, the magnitude of GM-CSF and MCP-1 induced arteriogenesis was reduced by approximately 40 % when ASA was co-administered; in contrast, Clopidogrel when used in the same model was neutral.

There is broad international agreement that patients with a generalized atherosclerosis and particularly patients suffering from PAD (who are at high risk for ischemic coronary and/or cerebral complications) should be treated with an antiaggregant. For pharmacoeconomic reasons the drug of choice normally is ASA.

However, following Höfer's results, ASA, although effectively preventing thrombotic complications, may hinder the arteriogenetic process required to normalize the physical capacity and QoL of PAD patients, a negative ASA effect which is not found with Clopidogrel.

Preliminary data in humans seem to support the hypothesis that in symptomatic stage II PAD patients Clopidogrel may be superior to ASA, a hypothesis which, in order to become conclusive, must be confirmed by the results of an evidence level 1 clinical trial.

(Literature at the Centre).

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for CD stability testing:

   * Patients of both sexes with subjectively reported initial claudication distances between 50 and 500 m
   * Patients with treadmill tested initial claudication distances between 50 and 400 m
   * History of intermittent claudication > 3 months
   * Established PAD diagnosis (ABI reference leg < 0.95 in non-diabetics, TBI reference leg < 0.70 in diabetics)
   * CLI ruled-out (ankle pressures > 50 mmHg (non diabetics), toe pressures > 30 mmHg (diabetics))
   * Stabilized treatment of concomitant diseases
2. Inclusion criteria for randomized treatment phase:

   * Patients of both sexes with treadmill tested initial claudication distances between 50 and 400 m
   * ICD variability during stability testing phase less than 25 %
   * History of intermittent claudication > 3 months
   * Established PAD diagnosis (ABI reference leg < 0.95 in non-diabetics, TBI reference leg < 0.70 in diabetics)
   * CLI ruled-out (ankle pressures > 50 mmHg (non diabetics), toe pressures > 30 mmHg (diabetics))
   * Stabilized treatment of concomitant diseases
   * Written informed consent

Exclusion Criteria:

* Treatment with oral anticoagulants (except those cases, where the parallel treatment with a platelet aggregation inhibitor (ASA, Clopidogrel) and an oral anticoagulant is medically indicated and justified)
* Lower extremity surgical reconstruction or PTA within the last 3 months
* Age < 45 years old (M), childbearing potential (F)
* Buerger's disease
* Clinically evident peripheral polyneuropathy (sensibility to vibration < 4/8, ATR not revocable)
* Presence of orthopedic, cardiac, pulmonary, or other concomitant diseases interfering with or preventing steady walking on a treadmill
* Clinically manifested congestive cardiac failure (NYHA class II - IV)
* Pretreatment with vasotherapeutics within the last 4 weeks prior to recruitment to the study without appropriate wash-out (> 5 half life times of the vasoactive drug)
* Consuming disease with life expectancy of less than 2 years
* Noncompliance of patient due to personality disorders or concomitant disease
* Known ASA or Clopidogrel intolerance
* Conditions requiring the regular intake of non-steroidal anti-inflammatory drugs
* Peptic ulcer within the previous 6 months
* History of GI or any other bleeding disorder within the previous 6 months

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Absolute claudication distance (ACD) change after prescription (Rx) | 3 Months

SECONDARY OUTCOMES:
Change in daily walking activity, quality of life (QoL), initial claudication distance (ICD) change after Rx | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kurt A Jaeger, MD, Prof, Principal Investigator — University Hospital, Basel, Switzerland; Ulrich Hoffmann, MD, Prof, Principal Investigator — University Hospital Munich (LMU)
Locations (16):
- Germany (6):
  - Evangelisches Krankenhaus Hubertus, Berlin
  - Dr. Doris Schulte, Berlin
  - Max Ratschow Klinik Darmstadt, Darmstadt
  - University Hospital Dresden, Dresden
  - Klinikum Karlsbad-Langensteinbach, Karlsbad
  - University Hospital Munich, Munich
- Switzerland (10):
  - University Hospital Basel Dpt. Angiology, Basel
  - Ospedale San Giovanni, Bellinzona
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Thurgau, Frauenfeld
  - University Hospital LAusanne, Lausanne
  - Kantonsspital Liestal, Liestal
  - Ospedale La Carita, Locarno
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

REFERENCES:
- [Derived] Singer E, Imfeld S, Staub D, Hoffmann U, Buschmann I, Labs KH, Jaeger KA. Effect of aspirin versus clopidogrel on walking exercise performance in intermittent claudication-a double-blind randomized multicenter trial. J Am Heart Assoc. 2012 Feb;1(1):51-6. doi: 10.1161/JAHA.111.000067. Epub 2012 Feb 20. PMID 23130118